CLINICAL TRIAL: NCT00735020
Title: A Phase I, Observer-Blind, Randomized, Single-Center Study to Evaluate Safety, Tolerability and Immunogenicity of a Bedside Mixing Combination of Two Adjuvanted Influenza Vaccines in Healthy Adults Aged 18 to 39 Years.
Brief Title: Study to Evaluate Safety, Tolerability and Immunogenicity of a Bedside Mixing Combination of Two Adjuvanted Influenza Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V104P1
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Influenza
Keywords: influenza; vaccine; adjuvants; flu
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: Adjuvanted Influenza Vaccine
- 2 (Active Comparator)
  Interventions: Biological: Influenza Vaccine

INTERVENTIONS:
Biological: Adjuvanted Influenza Vaccine — 1 dose of Adjuvanted Influenza Vaccine
  Arms: 1
Biological: Influenza Vaccine — 1 dose of Influenza Vaccine
  Arms: 2

SUMMARY:
This trial is designed to evaluate safety, tolerability and immunogenicity of a bedside mixing formulation of adjuvanted influenza vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 18 to 39 year old males and females who are in good health and have provided informed consent prior to enrollment

Exclusion Criteria:

* serious medical conditions
* allergies to vaccine components, including but not limited to egg/chicken products
* reduced immune function
* recent use of immunosuppressive therapy
* recent use of influenza vaccine

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Safety as measured through local and systemic reactions and efficacy (immunogenicity) as measured by antibody titers. | 36 Days

SECONDARY OUTCOMES:
To evaluate immunogenicity of a single IM injection of adjuvanted Influenza vaccine | 36 Days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- I.P.A.S., Ligornetto, Switzerland

REFERENCES:
- [Result] Della Cioppa G, Vesikari T, Sokal E, Lindert K, Nicolay U. Trivalent and quadrivalent MF59((R))-adjuvanted influenza vaccine in young children: a dose- and schedule-finding study. Vaccine. 2011 Nov 3;29(47):8696-704. doi: 10.1016/j.vaccine.2011.08.111. Epub 2011 Sep 9. PMID 21906647